CLINICAL TRIAL: NCT02458040
Title: Clinical Benefit of Genetic Biomarkers for Guiding Treatment Decisions in Oncology Drugs
Status: Withdrawn | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: BENEBIO01; PHRCK14-051 (Other Grant/Funding Number: Institut National du Cancer, France)
Record Dates: First submitted 2015-05-19; First posted 2015-05-29 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2015-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Biomarker-positive patients
  Interventions: Drug: Drug selected in the study
- Biomarker-negative patients
  Interventions: Drug: Drug selected in the study
- All patients
  Interventions: Drug: Drug selected in the study

INTERVENTIONS:
Drug: Drug selected in the study

SUMMARY:
This study is a meta-epidemiological study which aim is to quantify the clinical benefit of the biomarker-based strategy compared to conventional strategy across all drugs with such a strategy.

DETAILED DESCRIPTION:
Personalized medicine consist to differentially treat patients based on their individual characteristics (mainly genetics). It is of the most promising area of cancer research and cancer care. The label of more than 140 FDA- approved drugs mention a biomarker, the majority being indicated in oncology. However, it has also been suggested that the hopes of personalized medicine were not matched by evidence. Indeed, there is a threat that genetic biomarkers are used without evidence that this use translates in improved outcomes for patients, and the use of biomarkers is in need for thorough validation.

In a previous work the investigators showed that the mention of a pharmacogenomic biomarker in a drug label can have different meanings depending on the drug, and that oncology had higher proportion of required or recommended genetic testing compared to other therapeutic areas. Hence, the investigators will include only the drug-biomarker pairs with (i) required or recommended genetic testing, or (ii) with biomarker-based indication and (iii) with at least one indication in oncology.

ELIGIBILITY:
Inclusion Criteria:

* phase II or III randomized clinical trials
* including patients with one of the drug-biomarker-indication triplet studied
* evaluating treatment effect in biomarker-defined strata (either in biomarker-positive patients, in biomarker-negative patients or in both strata).
* reporting OS or PFS or DFS

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a systematic review. No patient will be directly included in this study, but the investigators will include clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 5 years

OTHER OUTCOMES:
Disease-Free Survival (DFS) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Hôtel Dieu, Paris, France

REFERENCES:
- [Background] Vivot A, Boutron I, Ravaud P, Porcher R. Guidance for pharmacogenomic biomarker testing in labels of FDA-approved drugs. Genet Med. 2015 Sep;17(9):733-8. doi: 10.1038/gim.2014.181. Epub 2014 Dec 18. PMID 25521333
- [Result] Vivot A, Boutron I, Beraud-Chaulet G, Zeitoun JD, Ravaud P, Porcher R. Evidence for Treatment-by-Biomarker interaction for FDA-approved Oncology Drugs with Required Pharmacogenomic Biomarker Testing. Sci Rep. 2017 Jul 31;7(1):6882. doi: 10.1038/s41598-017-07358-7. PMID 28761069